CLINICAL TRIAL: NCT01741493
Title: A Study in Healthy Adult Volunteers and Adult Subjects With Rheumatoid Arthritis to Evaluate the Safety, Tolerability, and Pharmacokinetics After Multiple Dosing of ABT-494
Brief Title: A Study in Healthy Adults and Adult Subjects With Rheumatoid Arthritis to Evaluate the Safety, Tolerability and Pharmacokinetics After Multiple Doses of ABT-494
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: M13-845
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Methotrexate; Tolerability; Pharmacokinetics; Safety; Tofacitinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib; tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (ABT-494) (Experimental): Multiple dosing of ABT-494 in healthy volunteers
  Interventions: Drug: ABT-494
- Rheumatoid Arthritis Patients (Experimental): Multiple dosing of ABT-494 in patients with rheumatoid arthritis
  Interventions: Drug: ABT-494
- No treatment (Placebo Comparator): Placebo administration in healthy volunteers and patients with rheumatoid arthritis
  Interventions: Drug: Placebo
- Healthy Volunteers (tofa) (Other): Multiple dosing of tofacitinib in healthy volunteers
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: ABT-494 — Oral administration of ABT-494 capsules
  Arms: Healthy Volunteers (ABT-494); Rheumatoid Arthritis Patients
Drug: Placebo — Oral administration of placebo capsules
  Arms: No treatment
Drug: Tofacitinib — Oral administration
  Arms: Healthy Volunteers (tofa)

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, multiple ascending dose study in healthy volunteers, multiple dose study in patients with rheumatoid arthritis and multiple dose study in healthy volunteers.

DETAILED DESCRIPTION:
To assess the safety, tolerability and pharmacokinetics of ABT-494 in healthy volunteers and in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Male and female subjects 18 to 55 years of age, inclusive.
* Subject is judged to be in good general health.

Rheumatoid Arthritis Patients:

* Male and female patients 18 to 75 years of age, inclusive.
* Subject has a diagnosis of rheumatoid arthritis for at least six months.
* Subject has been on methotrexate therapy for at least three months and on a stable dose for at least four weeks.

Exclusion Criteria:

* History or evidence of active or latent tuberculosis.
* History or significant allergic reaction to any drug.
* Use of known strong CYP3A and CYP2D6 inhibitors and CYP3A inducers within 21 days or within 5 half-lives of the respective medication, whichever is longer.
* Current or expected need for oral intake of at least 10 mg prednisone per day or equivalent corticosteroid therapy.
* History of acute inflammatory joint disease of different origin other than rheumatoid arthritis (rheumatoid arthritis patients).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with Adverse Events | From first dose up to 28 days after the last dose of study drug
Vital Signs | From first dose up to 28 days after the last dose of study drug
  Blood pressure, pulse rate and body temperature
Clinical Lab testing | From date of first dose up to 28 days after the last dose of study drug
  Hematology, Chemistry, and Urinalysis
Electrocardiogram (ECG) | Prior to first dose, during first dose interval, prior to last dose and until 24 hours post last dose
  ECGs done in triplicate; heart rate, PR interval, QT/QTc interval and QRS duration
Pharmacokinetics of ABT-494 | Prior to first dose up to 72 hours after the last dose of ABT-494
  Cmax, Tmax, AUC, elimination rate constant and half-life

SECONDARY OUTCOMES:
Pharmacokinetics of Methotrexate | Prior to first dose up to 48 hours after the last dose of methotrexate
  Cmax, Tmax, AUC, elimination rate constant and half-life

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jungerwirth, MD, Study Director — AbbVie
Locations (5):
- United States (5):
  - Site Reference ID/Investigator# 95817, Miami, Florida
  - Site Reference ID/Investigator# 95816, Cincinnati, Ohio
  - Site Reference ID/Investigator# 95815, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 92153, Austin, Texas
  - Site Reference ID/Investigator# 97177, Orem, Utah

REFERENCES:
- [Result] Mohamed MF, Camp HS, Jiang P, Padley RJ, Asatryan A, Othman AA. Pharmacokinetics, Safety and Tolerability of ABT-494, a Novel Selective JAK 1 Inhibitor, in Healthy Volunteers and Subjects with Rheumatoid Arthritis. Clin Pharmacokinet. 2016 Dec;55(12):1547-1558. doi: 10.1007/s40262-016-0419-y. PMID 27272171
- [Derived] Klunder B, Mohamed MF, Othman AA. Population Pharmacokinetics of Upadacitinib in Healthy Subjects and Subjects with Rheumatoid Arthritis: Analyses of Phase I and II Clinical Trials. Clin Pharmacokinet. 2018 Aug;57(8):977-988. doi: 10.1007/s40262-017-0605-6. PMID 29076110